CLINICAL TRIAL: NCT04694755
Title: An Exploratory Clinical Study on Reducing AECOPD of Chronic Respiratory Failure With COPD by Syndrome Differentiation
Brief Title: Treatment of CRF With Syndrome Differentiation of TCM
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Treatment of CRF with TCM
Record Dates: First submitted 2020-01-22; First posted 2021-01-05 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-08

CONDITIONS: Chronic Respiratory Failure
Keywords: COPD; Chronic respiratory failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Prescriptions

STUDY DESIGN:
Intervention Model Description: The experimental group was given TCM syndrome differentiation treatment granules, heart and lung qi deficiency was given invigorating heart and lung formula, lung and kidney qi deficiency was given invigorating kidney and protecting lung formula; the control group was given TCM syndrome differentiation treatment placebo.
Who Masked: Participant, Investigator
Masking Description: It is jointly completed by the person in charge of the project, the drug preparation personnel and the statistician, and the two-level blind method is adopted. Blinding at the first level: that is to say, blinding is set for experimental Chinese medicine. The test drug and the control drug shall be packed uniformly; the second level shall be provided with blindness, that is, the number of the test drug packaging box shall be provided with blindness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Heart lung qi deficiency syndrome placebo group (Placebo Comparator): Buyixinfei placebo was given.Tianjiang brand formula granules were used. One dose a day, two times orally, five days a week.
  Interventions: Drug: Placebo
- Deficiency of lung and Kidney Qi placebo group (Placebo Comparator): Tonifying kidney and protecting lung prescription placebo was given. Tianjiang brand granule was used as the drug, one dose a day, twice orally, five days a week.
  Interventions: Drug: Placebo
- Heart lung qi deficiency syndrome drugs group (Experimental): Buyixinfei formula was given. Tianjiang brand granule was used as the drug, one dose a day, twice orally, five days a week.
  Interventions: Drug: Traditional Chinese medicine prescription
- Deficiency of lung and Kidney Qi drugs group (Experimental): The prescription of invigorating the kidney and protecting the lung was given. The drug was Tianjiang brand granule, one dose a day, two times orally, five days a week
  Interventions: Drug: Traditional Chinese medicine prescription

INTERVENTIONS:
Drug: Placebo — On the basis of dextrin and bitter agent, 5% of the drug was used to prepare.Its appearance, weight, color and smell are basically the same as traditional Chinese medicine granule.Tianjiang brand formula granules, in line with GMP standards
  Other Names: Placebo for invigorating heart and lung; Tonifying kidney and protecting lung prescription placebo
  Arms: Deficiency of lung and Kidney Qi placebo group; Heart lung qi deficiency syndrome placebo group
Drug: Traditional Chinese medicine prescription — Tianjiang brand formula granules, in line with GMP standards
  Other Names: Tonic heart and lung prescription; Prescription for tonifying kidney and protecting lung
  Arms: Deficiency of lung and Kidney Qi drugs group; Heart lung qi deficiency syndrome drugs group

SUMMARY:
Taking the patients with chronic respiratory failure caused by COPD as the research object and the acute exacerbation of COPD as the main outcome index, the investigators hope to establish the syndrome differentiation and treatment scheme of COPD treated by traditional Chinese medicine, reduce the acute exacerbation of AECOPD, improve the clinical symptoms, improve the quality of life, reduce the mortality, preliminarily explore the mechanism of action, and lay the foundation for further research.

DETAILED DESCRIPTION:
Chronic respiratory failure of chronic obstructive pulmonary disease belongs to the category of "lung distention", "asthma syndrome", "dyspnea" and "phlegm drink" in traditional Chinese medicine. According to traditional Chinese medicine, the pathology of this disease is mainly the dysfunction of lung ventilation. The basic pathogenesis is that the viscera are repeatedly affected by evil, the lung qi is damaged due to long-term disease, the lung function is damaged, the air mechanism is blocked, the application is publicized, the phlegm is turbid, the blood stasis is inevitable for a long time, and the lung qi is further damaged. The main clinical manifestations are shortness of breath, wheezing, shortness of breath, superficial shortness of breath and "drama of wheezing when moving", which may be accompanied by cough, expectoration, chest tightness, palpitation, lips, purple darkness, swelling of floating limbs, etc. The treatment of chronic respiratory failure patients with COPD can be significantly improved clinical symptoms such as shortness of breath and wheezing, reduce the number of acute exacerbations of patients, but there is still a lack of high-level evidence-based medicine research. Therefore, this project puts forward the hypothesis that "syndrome differentiation therapy can reduce AECOPD of COPD".It is proposed to adopt a multicenter, randomized, double-blind, placebo-controlled trial design, taking the patients with chronic respiratory failure caused by chronic obstructive pulmonary disease as the research object. The patients who meet the inclusion criteria, are divided into heart lung qi deficiency and lung kidney qi deficiency according to syndrome differentiation. The participants are randomly divided into the experimental group of 60 cases and the control group of 60 cases. The control group is given placebo treatment, and the experimental group is given Chinese medicine granules. The patients were followed up for 26 weeks. The main outcome indicators include the number of times of acute exacerbation of COPD, and the secondary outcome indicators include all-cause mortality, severity of acute exacerbation of COPD, clinical symptoms, CCQ score of COPD clinical questionnaire, quality of life score, dyspnea score, 6MWD, arterial blood gas analysis index, incidence and use time of mechanical ventilation, use time of oxygen therapy, serology index, health and economy Learning indicators, safety indicators, etc. To establish the TCM treatment scheme of chronic respiratory failure of COPD, reduce the acute aggravation of AECOPD, improve the clinical symptoms, improve the quality of life, reduce the mortality rate, preliminarily explore the mechanism of action, and lay the foundation for further research.

ELIGIBILITY:
Inclusion criteria

1. patients who meet the diagnostic criteria of COPD in stable stage;
2. patients whose blood gas analysis meets PaO2 < 60mmhg and / or PaCO2 > 50mmhg in calm breathing at sea level;
3. patients whose syndrome differentiation meets the syndrome of heart lung qi deficiency and lung kidney qi deficiency;
4. patients whose age is ≥ 40 years and ≤ 80 years;
5. patients who are willing to receive treatment and sign the informed consent.

exclusion criteria:

1. chronic respiratory failure caused by bronchial asthma, bronchiectasis, cystic pulmonary fibrosis, lung cancer and other respiratory diseases;
2. acute aggravation of the original chronic respiratory failure;
3. patients with tumor, serious cardiovascular and cerebrovascular diseases (acute myocardial infarction, cardiac function level 3 and above, stroke, cerebral hemorrhage, etc.) and serious liver and kidney diseases (serious liver disease refers to liver cirrhosis, portal hypertension and varicose bleeding, and serious kidney disease includes dialysis and kidney transplantation) and other people who cannot participate in clinical research;
4. pregnant and lactating women;
5. patients with mental diseases and mental disorders;
6. those who are participating in clinical trials of other drugs, known to be allergic to treatment drugs.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of acute exacerbation | Up to week 52.
  It will be assessed by frequencies of AECOPD-related hospitalizations.
Duration of acute exacerbation | Up to week 52.
  Duration of acute exacerbation will be recorded.

SECONDARY OUTCOMES:
All-cause mortality | up to 52 weeks.
  The all-cause mortality will be calculated in each group at the end of the trial.
Dyspnea | Change from baseline mMRC scores at week 4, 13, 26, 39 and 52.
  Dyspnea will be assessed by modified Medical Research Council (mMRC) scores set up by American Thoracic Society. A score of 0-4 will be given according to the degree of immediate dyspnea. A higher score indicates a worse dyspnea.
COPD assessment test (CAT) | Change from baseline CAT scores at week 4, 13, 26, 39 and 52.
  CAT will be used to evaluate quality of life. A total score of 0-40 will be given with a higher score indicating a worse condition.
Clinical symptoms and Signs | Change from baseline clinical symptoms assessment questionnaire scores at week 4, 13, 26, 39 and 52.
  Assessment will be performed by clinical symptom assessment questionnaire. The clinical symptoms to be evaluated in this study include cough, expectoration, chest tightness, shortness of breath, wheezing and cyanosis. A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
Six-minute walking distance(6MWD) | Change from baseline 6MWD at week 4, 13, 26, 39 and 52
  6MWD will be applied to evaluate the exercise capacity. The higher values indicate the better exercise capacity.
CCQ | Change from baseline clinical symptom assessment questionnaire scores at week 4, 13, 26, 39 and 52.
  Clinical symptom assessment questionnaire of COPD (CCQ) will be used to assess symptom. There are 10 items with a score of 0-6 for each item. A higher value will indicate a worse symptom.
FEV1 | Change from baseline FEV1 at week 26 and 52.
  Forced expiratory volume in one second ( FEV1) will be applied to assess pulmonary function.
FVC | Change from baseline FVC at week 26 and 52.
  Forced vital capacity (FVC) will be applied to assess pulmonary function.
PaO2 | Change from baseline ABG at week 13, 26, 39 and 52.
  Partial pressure of oxygen (PaO2) will be applied to assess artery blood gas. PaO2≤60mmHg will indicatea the body is in a state of hypoxi.
PaCO2 | Change from baseline ABG at week 13, 26, 39 and 52.
  Partial pressure of carbon dioxide (PaCO2) will be applied to assess artery blood gas. PaCO2≥50mmHg will indicatea the body is in a state of carbon dioxide retention.
Duration of oxygen inhalation | Change from baseline Duration of oxygen inhalation at week 4, 13, 26, 39 and 52.
  Duration of oxygen inhalation will be used to evaluate quality of life. The longer the use, the worse the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Minghang Wang, doctor, Study Director — The First Affiliated Hospital of Henan University of Chinese Medicine